CLINICAL TRIAL: NCT05973279
Title: The Relationship Between Lower Limb Functionality, Knee Joint Position Sense, Balance and Falls in Haemiplegic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karabuk University (Other)
Collaborators: Bolu Izzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Fatma Hale Altınkaya, INVESTIGATOR, Karabuk University
Other Study IDs: KarabukUNI
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Haemiplegic Patients; Balance; Knee Joint Position Sensation; Lower Limb Functionality
Keywords: Proprioception; Joint Position Sense; Hemiplegia; Lower Limb Functionality; Balance; Fall
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemiplegic patients
  Interventions: Other: Tecno Body Prokin Isokinetic Balance System; Other: Restorative Therapies RT300 leg/arm/cor:; Other: CSMI (CYBEX) Humac Norm Isokinetic Test and Exercise System

INTERVENTIONS:
Other: Tecno Body Prokin Isokinetic Balance System — It provides objectively measurable data in static and dynamic balance measurements. The moving balance platform of the system, which is driven by air piston servo motors, can measure at a working angle of 15 degrees in all directions. The results can be monitored and recorded live on the screen on the device. From these data, each individual's static and dynamic balance score is obtained by summing the forward-backward standard deviation and right-left standard deviation.
Other: Restorative Therapies RT300 leg/arm/cor: — RT300 is a motorised treatment system. In general there are 3 systems; Passive therapy, Active therapy and a combination of active therapy with some assistance from the motor. The device can be used from a chair, wheelchair or bed and there are two variants that can be used separately; Leg system, Arm system. Electrodes placed on the skin over specific muscle groups are connected via a cable or wirelessly to the RT300. These are used to stimulate peripheral motor nerves, causing the muscles to work. The software of the SAGE controller unit of the RT300 monitors the treatment process, including the stimulation patterns sent to the arms or legs, and the operation of the ergometer motor to produce smooth cycling motion. Contraindicated in the presence of lower limb fractures or pregnancy.
Other: CSMI (CYBEX) Humac Norm Isokinetic Test and Exercise System — 22 isolated joint movement models, 4 resistance modes (isokinetic, isotonic, isometric and passive) and a large number of reports to meet the measurement and exercise needs of today's clinicians and researchers. The exercise modes of the device include; Continuous passive movement, multi-angle isometry, proprioception training, standard and eccentric focused isokinetic strengthening, deceleration training, dynamic isotonic training, strength training. Test modes of the device include; Proprioceptive, co-measured, standard isokinetic, concentric/eccentric isokinetic, intermittent stroke isokinetic test.

SUMMARY:
Stroke is defined as a neurological disorder attributed to acute focal damage of the central nervous system from a vascular cause, including cerebral infarction, intracerebral haemorrhage and subarachnoid haemorrhage. The World Health Organisation defines stroke as a focal and sometimes global impairment of cerebral function that lasts longer than 24 hours or ends in death, develops rapidly, has no demonstrable cause other than a vascular cause. Evaluation of muscle strength and balance ability of affected patients is critical for the recovery of lower extremity motor functions.

Proprioception encompasses various sensory perception modalities such as force, effort, movement and limb position. Impairment of sensory function in patients with haemiplegia can hinder the ability of muscles to recover during walking. Accurate and effective assessment of gait and balance functions and their subsequent improvement is one of the primary goals of stroke rehabilitation programmes. Studies comparing the effects of lower extremity functionality and knee joint position sense on balance and falls are available in various versions in the literature. However, there is no study in which 'Restorative Therapies RT300 leg/arm/cor' device was used to measure functionality, 'Humac Norm Isokinetic Machine' was used to measure knee joint position sense, and 'Tecno Body Prokin Isokinetic Balance System' was used to measure balance in a single simultaneous study. Therefore, the aim of this study was to investigate the relationship between lower limb functionality and knee joint position sense with balance and fall parameters in patients with hemiplegia using various devices.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age
* Volunteering to participate in the study

Exclusion Criteria:

* Hip and knee prosthesis
* Being diagnosed with vertigo
* Having a history of serious neurological diseases such as Parkinson's disease, multiple sclerosis except hemiplegia
* Having a previous operation for the lower limb
* Poor co-operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemiplegic patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Balance and knee joint position | First day
  Knee joint position sense is related to balance in haemiplegic patients.
Lower extremity functionality and balance | First day
  In haemiplegic patients, the level of lower extremity functionality is related to balance.
Falling and knee joint position | First day
  Knee joint position sense is associated with falls in haemiplegic patients.
Lower extremity functionality and falling | First day
  Lower extremity functionality is associated with falls in haemiplegic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Demirel, Study Director — Izzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Undecided